CLINICAL TRIAL: NCT06293378
Title: Safety and Effectiveness of Sulfasalazine in the Treatment of Liver Fibrosis/Cirrhosis.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Second Affiliated Hospital of Chongqing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Pengmingli
Record Dates: First submitted 2024-01-17; First posted 2024-03-05 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Cirrhosis, Liver; Fibrosis, Liver
MeSH Terms: conditions — Liver Cirrhosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Cohort A：Patients with PBC were treated with sulfasalazine (Experimental): PBC treatment group:
  1. PBC patients with poor response to UDCA after treatment: 30 patients continued to take UDCA 13-15mg/kg , 30 patients took UDCA 13-15mg/kg +SASP (0.5g orally three times a day), 30 patients took SASP (0.5g orally three times a day) for 12 months of follow-up observation. During 12 months of treatment, at the time of enrollment and the 1st/3rd/6th/9th/12th months, the liver function, fecal flora, liver fibrosis and immune related indexes were detected.
  2. Newly treated PBC patients: 30 patients took UDCA 13-15mg/kg and 30 patients took UDCA 13-15mg/kg +SASP (0.5g orally three times a day) for 12 months of follow-up observation. During 12 months of treatment, at the time of enrollment and the 1st/3rd/6th/9th/12th months, the liver function, fecal flora, liver fibrosis and immune related indexes were detected.
  Interventions: Drug: Sulfasalazine enteric-coated tablets
- Cohort B：Patients with HBV were treated with sulfasalazine (Experimental): Cohort B: 60 cases with hepatitis B cirrhosis were collected , 30 cases continued the current treatment(people with hepatitis B cirrhosis continue to take antivirals), and 30 patients were taking sulfasalazine for 12 months of follow-up observation. During 12 months of treatment, at the time of enrollment and the 1st/3rd/6th/9th/12th months, the liver function, fecal flora, liver fibrosis and immune related indexes were detected.
  Interventions: Drug: Sulfasalazine enteric-coated tablets
- Cohort C：Patients with HCV were treated with sulfasalazine (Experimental): Cohort C: 60 cases with hepatitis C cirrhosis were collected，30 cases continued the current treatment(people with hepatitis C cirrhosis continue to take antivirals), and30 patients were taking sulfasalazine for 12 months of follow-up observation. During 12 months of treatment, at the time of enrollment and the 1st/3rd/6th/9th/12th months, the liver function, fecal flora, liver fibrosis and immune related indexes were detected.
  Interventions: Drug: Sulfasalazine enteric-coated tablets
- Cohort D：Patients with alcoholic liver fibrosis/cirrhosis were treated with sulfasalazine (Experimental): 60 cases with alcoholic cirrhosis were collected , 30 cases continued the current treatment and 30 patients were taking sulfasalazine for 12 months of follow-up observation. During 12 months of treatment at the time of enrollment and the 1st/3rd/6th/9th/12th months, the liver function, fecal flora, liver fibrosis and immune related indexes were detected.
  Interventions: Drug: Sulfasalazine enteric-coated tablets

INTERVENTIONS:
Drug: Sulfasalazine enteric-coated tablets — Sulfasalazine enteric-coated tablets Cohort A: PBC treatment group: (1) PBC patients with poor response to UDCA after treatment: 30 patients continued to take UDCA(13-15mg/kg), 30 patients took UDCA(13-15mg/kg)+SASP (0.5g orally three times a day), 30 patients took SASP (0.5g orally three times a day) for 12 months of follow-up observation. During 12 months of treatment, at the time of enrollment and the 1st/3rd/6th/9th/12th months, the liver function, fecal flora, liver fibrosis and immune related indexes were detected. (2) Newly treated PBC patients: 30 patients took UDCA(13- 15mg/kg) and 30 patients took UDCA(13-15mg/kg)+SASP (0.5g orally three times a day) for 12 months of follow-up observation. During 12 months of treatment, at the time of enrollment and the 1st/3rd/6th/9th/12th months, the liver function, fecal flora, liver fibrosis and immune related indexes were detected.
  Arms: Cohort A：Patients with PBC were treated with sulfasalazine
Drug: Sulfasalazine enteric-coated tablets — Cohort B:60 cases with hepatitis B cirrhosis were collected from each group, 30 cases continued the current treatment, and 30 patients were taking SASP (0.5g orally three times a day) for 12 months of follow-up observation. During 12 months of treatment, at the time of enrollment and the 1st/3rd/6th/9th/12th months, the liver function, fecal flora, liver fibrosis and immune related indexes were detected.
  Arms: Cohort B：Patients with HBV were treated with sulfasalazine
Drug: Sulfasalazine enteric-coated tablets — Cohort C：Patients with HCV were treated with sulfasalazine Cohort C: 60 cases with hepatitis C cirrhosis were collected，30 cases continued the current treatment(people with hepatitis C cirrhosis continue to take antivirals), and30 patients were taking SASP (0.5g orally three times a day) for 12 months of follow-up observation. During 12 months of treatment, at the time of enrollment and the 1st/3rd/6th/9th/12th months, the liver function, fecal flora, liver fibrosis and immune related indexes were detected.
  Arms: Cohort C：Patients with HCV were treated with sulfasalazine
Drug: Sulfasalazine enteric-coated tablets — Cohort D：Patients with alcoholic liver fibrosis/cirrhosis were treated with sulfasalazine 60 cases with alcoholic cirrhosis were collected , 30 cases continued the current treatment and 30 patients were taking SASP (0.5g orally three times a day) for 12 months of follow-up observation. During 12 months of treatment, at the time of enrollment and the 1st/3rd/6th/9th/12th months, the liver function, fecal flora, liver fibrosis and immune related indexes were detected.
  Arms: Cohort D：Patients with alcoholic liver fibrosis/cirrhosis were treated with sulfasalazine

SUMMARY:
This is a controlled, observational clinical study initiated by investigators to investigate the efficacy and safety of sulfasalazine in the treatment of cirrhosis in patients with cirrhosis. Four cohorts were planned: primary biliary cirrhosis, hepatitis B and C cirrhosis, and alcoholic cirrhosis. The four groups were divided into experimental group and control group, and the experimental group: each group of patients was orally treated sulfasalazine for 12 months, taken three times a day, each time taking 0.5g. The control group did not take sulfasalazine. After 12 months, Observe changes in patients' biochemical and imaging indicators, liver stiffness values, fecal microbiota, and metabolites before and after the use of sulfasalazine.

DETAILED DESCRIPTION:
This study is a controlled and observational clinical study initiated by the investigators to study the efficacy and safety of sulfasalazine in the treatment of cirrhosis in patients with cirrhosis, and to observe changes in patients' biochemical and imaging indicators, liver stiffness values, fecal microbiota, and metabolites before and after the use of sulfasalazine.

Four cohorts were planned to be included in this study:

Cohort A: Differences in cirrhosis changes with the addition of sulfasalazine to UDCA in PBC patients with an inadequate response to UDCA and treatment-naïve PBC patients.

Cohort B: Differences in changes in cirrhosis in patients with viral hepatitis B cirrhosis compared with the addition of sulfasalazine to antiviral (if possible, the same antiviral) therapy.

Cohort C: Differences in changes in cirrhosis in patients with viral hepatitis C cirrhosis compared with the addition of sulfasalazine to antiviral (if possible, the same antiviral) therapy.

Cohort D: Differences in differences in changes in cirrhosis compared with sulfasalazine in patients with alcoholic hepatitis cirrhosis.

Treatment options:

1. Patients with PBC who did not respond adequately to UDCA: 30 patients with poor response to treated PBC continued to take UDCA, 30 patients with poor response to treated PBC received UDCA+SASP (0.5 g orally three times daily), and 30 patients with poor response received SASP (0.5 g orally three times daily) for 12 months and were followed up for 12 months.

   Treatment-naïve PBC patients: 30 treatment-naïve PBC patients took UDCA, and 30 treatment-naïve PBC patients took UDCA+SASP (0.5 g orally three times a day) for 12 months and followed up for 12 months.
2. Treatment group of hepatitis B (hepatitis C) viral liver cirrhosis: 60 patients with hepatitis B (hepatitis C) viral cirrhosis were collected (using the same dose of antiviral drugs), 30 patients with hepatitis B (hepatitis C) viral cirrhosis took antiviral drugs, and 30 patients with hepatitis B (hepatitis C) virus cirrhosis were treated with sulfasalazine (0.5g three times a day) on the basis of taking antiviral drugs, and follow-up observation was observed for 12 months.
3. Treatment group of alcoholic hepatitis cirrhosis: 60 patients with alcoholic cirrhosis were collected, 30 patients with alcoholic cirrhosis did not take antifibrotic drugs, 30 cases of alcoholic cirrhosis took sulfasalazine (0.5g three times a day), and follow-up observation was observed for 12 months.

ELIGIBILITY:
Inclusion Criteria:

1. Sign the informed consent form before the trial and be able to complete the study in accordance with the requirements of the trial protocol;
2. The age is 18~70 years old (including boundary value), the weight of male subjects is not less than 45 kg, and the weight of female subjects is not less than 40 kg. Body mass index (BMI) in the range of 18~32kg/m2 (including critical value);
3. Enrolled patients also need to meet:

A:Patients with PBC cirrhosis PBC patients who have been treated and show an inadequate response to UDCA：(1) according to the biochemical response criteria for 2021 PBC, Enrolled patients need to meet the criteria of ALP ≥1.67 × ULN as a poor biochemical response to UDCA after 12 months of UDCA treatment; (2) meeting the diagnostic criteria for primary cholangitis (PBC) , i.e. meeting at least two of the following criteria: 1.indicators of cholestasis such as elevated Alkaline phosphatase; 2.Anti-mitochondrial antibody AMA or AMA-m2 positive, or if AMA negative, PBC-specific antibodies (anti-GP210 Andor anti-SP100) positive .3 liver biopsy consistent with PBC; Patients with newly diagnosed primary cholangitis (PBC-RRB- met the diagnostic criteria of at least two of the following): 1.indicators of cholestasis such as elevated Alkaline phosphatase; 2.Anti-mitochondrial antibody AMA or AMA-m2 positive, or if AMA negative, PBC-specific antibodies (anti-GP210 Andor anti-SP100) positive 3. liver biopsy consistent with PBC; B:Patients with hepatitis B cirrhosis Diagnosis of hepatitis B cirrhosis based on clinical history, histology or imaging.

C:Patients with hepatitis C cirrhosis Diagnosis of hepatitis C cirrhosis based on clinical history, histology or imaging.

D:Alcoholic hepatitis cirrhosis Diagnosis of alcoholic cirrhosis based on clinical history, histology, or imaging.

Exclusion Criteria:

1. Those who have a history of allergies in the past, or the investigator suspects that they are allergic to the active ingredients of the drug or their excipients under study;
2. Allergy to sulfasalazine and its metabolites, sulfonamides or salicylic acid;
3. Patients with intestinal obstruction or urinary tract obstruction;
4. Patients with porphyria, such as sulfonamides, have been reported to cause acute attacks.
5. Acute and chronic liver disease with clinical significance caused by infections other than HBV, HCV, PBC, and alcoholic liver disease;
6. Primary liver cancer; alpha-fetoprotein (AFP) greater than 50 ug/L or imaging suggests malignant liver mass; Those with other malignancies or a history of other malignancies in the 5 years prior to screening (except for complete remission of malignant tumors after treatment and no additional medical or surgical intervention within 3 years prior to screening);
7. The investigator judged that there is impaired gastrointestinal function or gastrointestinal diseases that may affect the absorption of oral drugs, such as severe gastric ulcer, erosive gastritis, partial gastrectomy, and persistent >Grade 2 gastrointestinal symptoms (e.g., nausea, vomiting, or diarrhoea);
8. Serious diseases of circulatory, respiratory, urinary, blood, metabolic, immune, psychiatric, neurological, renal and other systems;
9. Those who have had major trauma or undergone major surgery within 3 months before screening; or those who plan to undergo surgery during the study;
10. Donated blood or lost blood ≥ 400mL within 3 months before screening, or received blood transfusion; or ≥ blood donation or blood loss within 1 month prior to screening 200mL；
11. Those who are positive for AIDS antigen/antibody, positive for Treponema pallidum antibody and positive RPR test;
12. History of drug dependence or drug abuse within 1 year prior to screening;
13. Participate in clinical trials of other investigational drugs or medical devices within 3 months before screening, and take experimental drugs or use them Those who have medical devices;
14. Those who have a positive pregnancy test during lactation or screening, or who have fertility requirements in the past two years;
15. Subjects who the investigator believes have other factors that are not suitable to participate in this trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2028-10-10 (Estimated); Study Completion 2028-10-10 (Estimated)

PRIMARY OUTCOMES:
Hepatic fibrosis | baseline，1,3,6,9,12 months after treatment and 1 month after the end of treatment.
  The changes of liver fibrosis
Serum alkaline phosphatase (ALP) | baseline,1,3,6,9,12 months after treatment and 1 month after the end of treatment.
  Serum alkaline phosphatase (ALP) level
Serum γ-glutamyl transpeptidase (GGT) | baseline,1,3,6,9,12 months after treatment and 1 month after the end of treatment.
  Serum γ-glutamyl transpeptidase (GGT) level
Serum bilirubin | baseline,1,3,6,9,12 months after treatment and 1 month after the end of treatment.
  Serum bilirubin level
Serum bile acids | baseline,1,3,6,9,12 months after treatment and 1 month after the end of treatment.
  Serum bile acids level
Serum aspartate aminotransferase(AST) | baseline,1,3,6,9,12 months after treatment and 1 month after the end of treatment.
  Serum aspartate aminotransferase(AST) level
Serum alanine aminotransferase (ALT) | baseline,1,3,6,9,12 months after treatment and 1 month after the end of treatment.
  Serum alanine aminotransferase (ALT) level

SECONDARY OUTCOMES:
The gut microbiota and metabolites. | baseline,1,3,6,9,12 months after treatment and 1 month after the end of treatment.
  The levels of changes in gut microbiota and metabolites.

OTHER OUTCOMES:
Changes in immune cells | baseline,1,3,6,9,12 months after treatment and 1 month after the end of treatment.
  Th1 cells (CD3 + CD4 + IFN-γ +) , Th2 cells (CD3 + CD4 + IL-4 +) , Th17 cells (CD3 + CD4 + IL-17 +) , Treg cells (CD3 + CD4 + CD25 + CD127low) ,Tfh cells (CD3+CD4+CXCR5+CD127highCD25low), Tfh1 cells (CXCR3 + CCR6- on the basis of Tfh) , Tfh2 cells (CXCR3-CCR6- on the basis of Tfh) , Tfh17 cells (CXCR3-CCR6+ on the basis of Tfh) , Tfr cells (CD4+CXCR5+CD127lowCD25high)，activated CD8 + T cells (CD3 + CD8 + CD38 +) , B cells（CD3-CD19+），B regulatory cells（CD3-CD19 + CD24highCD38), Plasma cells(CD20lowCD27highCD38high based on B cells ).

CONTACTS AND LOCATIONS:
Overall Officials: Mingli Peng, Doctor, Study Chair — The Second Affiliated Hospital of Chongqing Medical University; Yinghua Lan, Doctor, Study Chair — Doctor
Locations (2):
- China (2):
  - Chongqing Medical University, Chongqing, Chongqing Municipality
  - Chongqing, Chongqing, Chongqing Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Gulamhusein AF, Hirschfield GM. Primary biliary cholangitis: pathogenesis and therapeutic opportunities. Nat Rev Gastroenterol Hepatol. 2020 Feb;17(2):93-110. doi: 10.1038/s41575-019-0226-7. Epub 2019 Dec 9. PMID 31819247
- [Result] Lv T, Chen S, Li M, Zhang D, Kong Y, Jia J. Regional variation and temporal trend of primary biliary cholangitis epidemiology: A systematic review and meta-analysis. J Gastroenterol Hepatol. 2021 Jun;36(6):1423-1434. doi: 10.1111/jgh.15329. Epub 2020 Dec 6. PMID 33141955
- [Result] Lindor KD, Bowlus CL, Boyer J, Levy C, Mayo M. Primary biliary cholangitis: 2021 practice guidance update from the American Association for the Study of Liver Diseases. Hepatology. 2022 Apr;75(4):1012-1013. doi: 10.1002/hep.32117. Epub 2021 Dec 20. No abstract available. PMID 34431119